CLINICAL TRIAL: NCT06719752
Title: ASSESSING the ACUTE EFFECTS of DIAGONAL MOBILIZATION on STATIC and DYNAMIC BALANCE in YOUNG FOOTBALL PLAYERS: a RANDOMIZED DOUBLE-BLIND STUDY
Brief Title: Assessing the Acute Effects of Diagonal Mobilization
Acronym: Manual Therapy
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KB/392/2023
Record Dates: First submitted 2024-11-30; First posted 2024-12-06 (Actual); Last update posted 2025-02-25 (Actual); Status verified 2025-02

CONDITIONS: Aged 14 to 16; Play Football Regularly
Keywords: soccer; musculoskeletal manipulations; postural balance; biomechanics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Assessing the acute effects of mobilization (Active Comparator): Participants will undergo an active intervention consisting of passive mobilization of rhythmic gliding.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo intervention; the therapy will mimic exceptional mobilization.

SUMMARY:
Investigating the acute effects of mobilization on these parameters offers innovative insights for the practitioner community and sheds light on the strategy's potential effectiveness in mitigating injury risk. Therefore, this study aims to assess the immediate effects of mobilization on static and dynamic balance in young male and female soccer players using a randomized, double-blinded study design.

DETAILED DESCRIPTION:
Participants underwent assessment twice: once before the intervention and again afterward. Tests included the single leg lend and hold test and the single leg standing test, measured using force plates.

ELIGIBILITY:
Inclusion Criteria:

* age between 14 to 16 years old, with regular soccer practice;
* absence of lower limb and lumbar spine surgery or injuries within the last 6 months (hip, knee, ankle), no current pain in the hip, knee, or ankle joints, no hypermobility of the lower limb joints, and no history of neurological or connective tissue disorders;
* availability for both assessment time points

Exclusion Criteria:

-

Ages: 14 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2025-02-25 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Single leg standing | 2-3 seconds
  Participants will initiate the evaluation by standing on force plates (ForceDecks, VALD, Brisbane, Australia) in a standard standing posture.

CONTACTS AND LOCATIONS:
Locations (1):
- AZS Central Academic Sports Center in Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Studnicki R, Taraszkiewicz M, Hansdorfer-Korzon R, Kawczynski A. Assessing the acute effects of diagonal mobilization on static and dynamic balance in young football players: a randomized double-blind study. BMC Sports Sci Med Rehabil. 2025 Jul 2;17(1):164. doi: 10.1186/s13102-025-01212-4. PMID 40604994